CLINICAL TRIAL: NCT04842747
Title: Phase 3, Randomized, Placebo-Controlled, Efficacy and Safety Study of VERU-111 for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) in Patients at High Risk for Acute Respiratory Distress Syndrome (ARDS).
Brief Title: VERU-111 in the Treatment of SARS-Cov-2 Infection by Assessing Its Effect on the Proportion of Patients Who Die on Study
Acronym: VERU-111
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Veru Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V3011902
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: SARS-CoV Infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — sabizabulin

STUDY DESIGN:
Intervention Model Description: Subjects in the VERU-111 treatment groups will receive standard of care, plus oral daily VERU-111 9mg for 21 days or until released from hospital. Subjects in the Placebo treatment group will receive standard of care, plus a placebo capsule for 21 days or until released from hospital.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be a randomized, double-blind, placebo-controlled study. Randomization will be stratified by baseline WHO Ordinal Scale score of 4,5 and 6 such that subjects with a WHO Ordinal Scale of 4, 5 and 6 at screening are approximately equally distributed between the treatment groups. An emergency code break will be available to the investigator / pharmacist / investigational drug storage manager. This code break option in IWRS may only be disclosed in emergency situations when the identity of the trial drug must be known to the investigator in order to provide appropriate medical treatment or if required to assure safety of trial participants. If the code break for a patient is opened, the sponsor and CRO will be informed immediately via IWRS notification. The reason for the IWRS unblinding of the subject must be documented on the appropriate eCRF page along with the date and the initials of the person who broke the code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 9mg of VERU-111 Oral daily (Experimental): 9mg of VERU-111
  Interventions: Drug: VERU-111
- Placebo Capsule once daily (No Intervention): Subjects in the Placebo treatment group will receive standard of care, plus a placebo capsule for 21 days or until released from hospital.

INTERVENTIONS:
Drug: VERU-111 — Subjects in the VERU-111 treatment groups will receive standard of care, plus oral daily VERU-111 9mg for 21 days or until released from hospital.
  Other Names: Sabizabulin
  Arms: 9mg of VERU-111 Oral daily

SUMMARY:
To demonstrate the efficacy of VERU-111 in the treatment of SARS-Cov-2 Infection by assessing its effect on the proportion of patients who die on study (prior to Day 60).

DETAILED DESCRIPTION:
This study is a multicenter, randomized, placebo-control, efficacy and safety study of VERU-111 for the treatment of COVID-19. Subjects will receive either 9mg of VERU-111 or matching placebo orally or through nasogastric tube daily for up to 21 days or until the subject is discharged from the hospital, whichever comes first. The primary efficacy endpoint of the study will be the proportion of subjects that die prior to Day 60.The total study duration for a subject from screening to follow up visit is planned to be 62 days. In addition to the safety of VERU-111, an evaluation of the efficacy of VERU-111 on SARS-CoV-2 (COVID-19) compared to the placebo control will be evaluated as part of the Independent Data Monitoring Committee (IDMC).

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent from the subject or the subject's Legally Authorized Representative (LAR)
* Aged ≥18 years
* Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) infection confirmed by polymerase chain reaction (PCR) test
* Patients with a WHO Ordinal Scale for Clinical Improvement score of 4 at high risk for ARDS, must have at least one of the known comorbidities for being at high risk, such as, Asthma (moderate to severe), Chronic Lung Disease, Diabetes, Hypertension, Severe Obesity (BMI ≥40), 65 years of age or older, primarily reside in a nursing home or long-term care facility, or immunocompromised and patients with a WHO Ordinal Scale for Clinical Improvement score of 5 or 6 regardless of presence of comorbidities.
* WHO Ordinal Scale for Clinical Improvement score of 4 (Oxygen by mask or nasal prongs), 5 (Non-invasive ventilation or high-flow oxygen) or 6 (Intubation and mechanical ventilation)
* Peripheral capillary oxygen saturation (SpO2) ≤ 94% on room air at screening. If patient is on oxygen therapy at the time of presentation for screening and the SpO2 levels were ≤94% prior to introduction to oxygen therapy with proper documentation example EMT notes or ER/ED notes, then the patient is considered to have met this inclusion criterion. If patient is on oxygen therapy at the time of presentation for screening and the SpO2 levels prior to introduction to oxygen therapy are unknown, the patient may be considered to have met this inclusion criterion if oxygen therapy is removed and the SpO2 levels fall to ≤94%, then the patient is considered to have met this inclusion criterion. However, removal of the oxygen therapy should only be done if it is considered medically reasonable
* Subjects must agree to follow doctor's recommendation for oxygen supplementation
* Subjects must agree to use acceptable methods of contraception:

  * If female of childbearing potential or a male subject's partner could become pregnant, use acceptable methods of contraception from the time of the first administration of study medication until 6months following administration of the last dose of study medication. Acceptable methods of contraception are as follows: Condom with spermicidal foam/gel/film/cream/suppository [i.e., barrier method of contraception], surgical sterilization (vasectomy with documentation of azospermia) and a barrier method {condom used with spermicidal foam/gel/film/cream/suppository}, the female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or subdermal implants and a barrier method (condom used with spermicidal foam/gel/film/cream/suppository)
  * If the female partner of a male subject has undergone documented tuballigation (female sterilization), a barrier method (condom used with spermicidal foam/gel/film/cream/suppository)should also be used
  * If female partner of a male subject has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS),a barrier method (condom with spermicidal foam/gel/film/cream/suppository)should also be used
* Subject is willing to comply with the requirements of the protocol through the end of the study

Exclusion Criteria:

* Known hypersensitivity or allergy to colchicine
* Pregnant or currently breast feeding
* Participation in any other clinical trial of an experimental treatment for COVID- 19. Convalescent plasma, dexamethasone and remdesivir are allowed in this study.
* Concurrent treatment with other experimental agents with actual or possible direct acting antiviral activity against COVID-19is prohibited <24 hours prior to study drug dosing(except standard of care). Remdesivir, dexamethasone and convalescent plasma are allowed in the study.
* Requiring ventilation + additional organ support - pressors, RRT, ECMO(WHO Ordinal Scale for Clinical Improvement - Score of 7). NOTE: short term (PRN) use of pressors is allowed
* Alanine Aminotransferase (ALT) or aspartate aminotransferase(AST) >3X upper limit of normal (ULN)
* Total bilirubin > ULN
* Creatinine clearance < 60 mL/min
* Documented medical history of liver disease, including but not limited to, prior diagnosis of hepatitis of any etiology, cirrhosis, portal hypertension, or confirmed or suspected esophageal varices
* Moderate to severe renal impairment
* Hepatic impairment
* History of hepatitis - (Hepatitis B and C) NOTE: treated and controlled hepatitis C is allowed
* Any comorbid disease or condition (medical or surgical) which might compromise the hematologic, cardiovascular, endocrine, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk
* Participants must agree to refrain from prolonged exposure to the sun or agree to use at least SPF 50 on all exposed skin and protective clothing during prolonged sun exposure throughout participation in this study and/or treatment with VERU-111

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barnette, Study Chair — Veru Inc.
Locations (58):
- United States (21):
  - Honor Health, Scottsdale, Arizona
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - Velocity Clinical Research, Chula Vista, California
  - Velocity Clinical Research - San Diego, La Mesa, California
  - Westchester General Hospital, Research Department, Miami, Florida
  - James A. Haley Veterans Hospital, Tampa, Florida
  - Wellstar Research Institute, Marietta, Georgia
  - Benchmark Research, Covington, Louisiana
  - Methodist Hospital, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Holy Name Medical Center, Institute for Clinical Research, Teaneck, New Jersey
  - Inspira Medical Center, Vineland, New Jersey
  - University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - The Stern Cardiovascular Foundation, Inc., Germantown, Tennessee
  - Regional One Health, Memphis, Tennessee
  - North Knoxville Medical Center, Powell, Tennessee
  - HD Research (Memorial Hermann - Memorial City Medical Center), Houston, Texas
  - HD Research (Memorial Hermann Southeast Hospital), Houston, Texas
  - Clinical Trial Network, Houston, Texas
- Argentina (5):
  - Hospital De Alta Compleijdad Cuenca Alta Nestor Kirchner, Buenos Aires
  - Hospital del Bicentenario de Esteban Echeverría, Buenos Aires
  - Center Sagrado Corazon, Buenos Aires
  - Sanatorio Güemes, Buenos Aires
  - Hospital De Infecciosas "Dr. Francisco Javier Muniz", Buenos Aires
- Brazil (15):
  - Fundacao Pio XII - Hospital de Amor de Barretos, Barretos, São Paulo
  - Hospital PUC Campinas, Campinas, São Paulo
  - Faculdade de Medicina de Botucatu - UNESP, Botucatu
  - Hospital Universitário São Francisco na Providencia de Deus, Bragança Paulista
  - IPECC (Instituto De Pesquisa Clínica de Campinas), Campinas
  - Sociedade Hospital Angelina Caron, Campinas
  - Santa Casa de Curitiba, Curitiba
  - Complexo Hospitalar de Niteroi, Niterói
  - Hospital de Clínicas de Porto Alegre - Infectologia - Centro de Pesquisa Clínica, Porto Alegre
  - Hospital Sao Luca Da PUCRS, Porto Alegre
  - Hospital Universitario Cementino Fraga Filho, Rio de Janeiro
  - IDOR - D'Or Institute for Research and Education, São Paulo
  - Incor - Instituto do Coração do Hospital das Clínicas da FMUSP, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São Paulo
  - Hospital Miguel Soeiro Sorocaba, Sorocaba
- Bulgaria (9):
  - MHAT Blagoevgrad AD Department of Infectious Diseases, Blagoevgrad
  - Multiprofile Hospital for Active Treatment - Haskovo, Department of Infectious Diseases, Haskovo
  - Multiprofile Hospital for Active Treatment - Dr. Atanas Dafovski AD, Kardzhali, Department of Pneumology and Phthisiatry, Dept. of Pneumology & Phthisiatry, Kardzhali
  - Specialized hospital for active treatment of pulmonary diseases -Pernik EOOD, Pernik, Pernik
  - University Multiprofile Hospital for Active Treatment "Pulmed" OOD Plovid Rheumatology, Plovdiv
  - MHAT Bratan Shukerov,Pulmonology Department, Smolyan
  - University Multiprofile Hospital for Active Treatment "Tsaritsa Yoanna-ISUL" EAD, Sofia,, Sofia
  - Multiprofile Hospital for Active Treatment and Emergency Medicine, Sofia
  - University Multiprofile Hospital for Active Treatment "Professor Doctor Stoyan Kirkovich" AD, Stara Zagora, Clinic of Anaestheology and intensive care, Stara Zagora
- Colombia (5):
  - Fundación Hospital Universidad del Norte (Barranquilla), Atlántico
  - Clinica de la Costa (Barranquilla), Barranquilla
  - Fundación Cardioinfantil-Instituto de Cardiología, Bogotá
  - Centro Medico Imbanaco de Cali S.A, Cali
  - Sociedad Medica Rionegro- Clínica Somer (Rionegro), Rionegro
- Mexico (3):
  - Unidad Médica para la Salud Integral (UMSI), San Nicolás de los Garza, Nuevo León
  - Hospital General de Culiacán, Culiacán
  - Hospital General de Occidente, Zapopan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barnette KG, Gordon MS, Rodriguez D, Bird TG, Skolnick A, Schnaus M, Skarda PK, Lobo S, Sprinz E, Arabadzhiev G, Kalaydzhiev P, Steiner M. Oral Sabizabulin for High-Risk, Hospitalized Adults with Covid-19: Interim Analysis. NEJM Evid. 2022 Sep;1(9):EVIDoa2200145. doi: 10.1056/EVIDoa2200145. Epub 2022 Jul 6. PMID 38319812

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 9mg of VERU-111 Oral Daily | Placebo Capsule Once Daily
Started | 134 | 70
Completed | 125 | 66
Not Completed | 9 | 4
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Subject refused all care decision was made to withdraw subject.No study IP given.IRB was consulted . | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 9mg of VERU-111 Oral Daily | Placebo Capsule Once Daily | Total
Number analyzed (Participants) | 134 | 70 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (14.14) | 62.7 (13.90) | 61.8 (14.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 26 | 70
  Male | 90 | 44 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 28 | 86
  Not Hispanic or Latino | 76 | 42 | 118
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 114 | 64 | 178
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  North America | 48 | 26 | 74
  South America | 55 | 27 | 82
  Europe | 31 | 17 | 48

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Sabizabulin in the Treatment of SARS-CoV-2 Infection by Assessing Its Effect on the Proportion of Patients Who Died on Study.
Description: Efficacy of VERU-111 in the treatment of SARS-Cov- 2 Infection by assessing its effect on the proportion of patients who die on study (prior to Day 60).
Time Frame: Day 60
Population: Intent to treat population of 204
Measure: Count of Participants; unit: Participants
Arm/Group | 9mg of VERU-111 Oral Daily | Placebo Capsule Once Daily
Number analyzed (Participants) | 134 | 70
Participants | 25 | 27

2. Secondary Outcome: The Proportion of Subjects That Are Alive Without Respiratory Failure at Day 15, Day 22 and Day 29.
Description: The proportion of subjects that are alive without respiratory failure at Day 15, Day 22 and Day 29. Respiratory failure is defined as endotracheal intubation and mechanical ventilation, extracorporeal membrane oxygenation, high-flow nasal cannula oxygen delivery, noninvasive positive pressure ventilation, clinical diagnosis of respiratory failure with initiation of none of these measures only when clinical decision making is driven solely by resource limitation.
Time Frame: Day 15, Day 22, Day 29
Population: Responders are subjects who are alive without respiratory failure at Day 15, Day 22 and Day 29.
Measure: Count of Participants; unit: Participants
Arm/Group | 9mg of VERU-111 Oral Daily | Placebo Capsule Once Daily
Number analyzed (Participants) | 134 | 70
Participants
  Day 15 | 94 | 40
  Day 22 | 96 | 39
  Day 29 | 96 | 38

ADVERSE EVENTS:
Time Frame: 60 Days
Description: Per protocol adverse events were captured from first dose thru day 60, resulting in this analysis to be the safety population of 199.
Arm/Group | 9mg of VERU-111 Oral Daily | Placebo Capsule Once Daily
All-Cause Mortality (participants affected / at risk) | 25/134 | 27/70
Serious Adverse Events (participants affected / at risk) | 38/130 | 32/69
Other Adverse Events (participants affected / at risk) | 82/130 | 54/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 9mg of VERU-111 Oral Daily (N=130) | Placebo Capsule Once Daily (N=69)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 3 (4)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Mydriasis (Eye disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2)
Procedural failure (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acinetobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Burkholderia cepacia complex infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (6) | 4 (5)
Pneumonia acinetobacter (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 4 (5) | 2 (2)
Sepsis Shock (Infections and infestations) | 2 (2) | 5 (5)
Severe acute respiratory syndrome (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure like phenomena (Nervous system disorders) | 1 (1) | 0 (0)
Stroke in evolution (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 6 (6)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 14 (14)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 9mg of VERU-111 Oral Daily (N=130) | Placebo Capsule Once Daily (N=69)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 5 (5)
Bradycardia (Cardiac disorders) | 6 (7) | 5 (5)
Constipation (Gastrointestinal disorders) | 9 (9) | 6 (10)
Pneumonia (Infections and infestations) | 8 (12) | 9 (12)
Septic shock (Infections and infestations) | 2 (2) | 5 (5)
Urinary tract infection (Infections and infestations) | 8 (8) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (6) | 6 (7)
Hypernatremia (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 6 (7) | 5 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 4 (5)
Anxiety (Psychiatric disorders) | 4 (5) | 4 (4)
Delirium (Psychiatric disorders) | 5 (5) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 11 (11) | 8 (8)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 14 (14)
Hypotension (Vascular disorders) | 5 (9) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT04842747/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT04842747/SAP_001.pdf